CLINICAL TRIAL: NCT02414425
Title: Effect And Tolerance of Botulinum A Toxin Rectal Injections on Fecal Incontinence
Acronym: FI_TOXIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/008/HP; 2014-003650-14 (EudraCT Number)
Record Dates: First submitted 2015-04-01; First posted 2015-04-10 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Botulinum Toxin A; Rectal injection
MeSH Terms: conditions — Fecal Incontinence | interventions — Proctoscopy; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectal Injection of Botulinum toxin A (Experimental): Botulinum toxin A will be injected during rectoscopy for patient with rectal incontinence.
  Anorectal manometry will be performed for evaluation of efficacy of experimental drug
  Interventions: Procedure: Rectoscopy; Procedure: Anorectal manometry; Drug: Botulinum toxin A or physiologic serum injection
- Rectal Injection of physiologic serum (Placebo Comparator): physiologic serum will be injected during rectoscopy for patient with rectal incontinence.
  Anorectal manometry will be performed for evaluation of efficacy of placebo
  Interventions: Procedure: Rectoscopy; Procedure: Anorectal manometry; Drug: Botulinum toxin A or physiologic serum injection

INTERVENTIONS:
Procedure: Rectoscopy — A rectoscopy will be performed for Botulinum toxin A or physiologic serum injection
Procedure: Anorectal manometry — Anorectal manometry will be performed to evaluate efficacy of Botulinum toxin A or physiologic serum rectal injection
Drug: Botulinum toxin A or physiologic serum injection — Botulinum toxin A or physiologic serum injection is performed during rectoscopy

SUMMARY:
Fecal incontinence is a frequent pathology which concerns 10% of the general population and severely alters patients quality of life. The cost of urinary and faecal incontinence has been estimated to be $16 billions a year. Several treatments exist depending on the aetiology of the faecal incontinence: medical treatments, biofeedback and sacral nerve stimulation. Nevertheless, these treatments are not always effective (50-70% of success) and are not without side effects, particularly the sacral nerve stimulation (pain, infection, electrode displacement..).

The intravesical injections of botulinum toxin have been used for several years for the treatment of urinary incontinence with overactive bladder. Several randomized trials have demonstrated the efficacy of these injections in patients with neurological disorders and overactive bladder, as well as in idiopathic overactive bladder. The toxin injections in the detrusor muscle increase the compliance and the bladder capacity and delay the initial appearance of detrusor uninhibited contraction. Furthermore, botulinum toxin decreases the urinary urgency. It maybe secondary to the reduction of the amplitude of the detrusor uninhibited contraction as well as to a direct effect of toxin on sensory pelvic nerve afferents.

The botulinum toxin should play a role on motor afferents as well as on the sensory function of efferent nerves.

The hypothesis is to demonstrate a decrease of active faecal incontinence and/or urgency episodes with improvement in quality of life, without any major side effects, in the patients included in this study. Nevertheless, the benefit of toxin injections are known to be temporary because of nerve re-growth. If we obtain similar results for fecal incontinence, it would be possible to schedule one to two injections a year because of the limited side-effects and invasiveness of the rectal injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one episode of active Fecal Incontinence and /or urgency per week;
* Patients with Fecal Incontinence for at least 3 months;
* Patients with Fecal Incontinence refractory to conventional treatment (medical and biofeedback);
* Patients having read the information letter and signed informed consent;
* Patients with medical insurance.

Exclusion Criteria:

* Patients younger than 18 years old;
* Pregnant or breast-feeding women or women without effective contraception and of age to procreate;
* Exclusive passive Fecal Incontinence;
* Fecal Incontinence secondary to anorectal malformation, post-surgery, anorectal organic disease (cancer, inflammatory bowel disease, post-radiotherapy etc.), constipation, an anal sphincter lesion which could be repaired as a first step, a rectal prolapse (the inclusion in the study is possible if Fecal Incontinence persists after rectopexy, a neurological disease with rapid progress ( stable neurological status is needed for at least 6 months);
* Patients under guardianship.
* Known Hypersensibility to botulinum toxin;
* Neuromuscular junction pathology (myasthenia, Lambert-Eaton syndrome);
* Anesthesia performed less than 1 month previously;
* Association with antibiotics
* Neurological pathology such as polyradiculoneuropathy;
* Dysphagia, pneumopathy secondary to dysphagia;
* Botulinum toxin injections during the 3 months before the beginning of the study;
* Known Hypersensitivity to albumin;
* History of inhalation pneumopathy.
* Rectoscopy impossible (anal stenosis for example);
* Anti-coagulant or anti-platelet drug or hemostasis disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Number of active fecaI incontinence episodes per week | 1 Month
  The number of fecaI incontinence episodes is evaluated using a bowel diary
Change from baseline in the Number of urgencies episodes per week | 1 Month
  The number of urgencies episodes is evaluated using a bowel diary

SECONDARY OUTCOMES:
Number of Adverse Events | 6 Months
  Imputability of Adverse events is evaluated by investigator
Number of Adverse Events | 1 Month
  Imputability of Adverse events is evaluated by investigator
Number of Adverse Events | 3 Months
  Imputability of Adverse events is evaluated by investigator
Change from baseline in the severity of fecal incontinence | 6 Months
  The severity of fecal incontinence is evaluated using Cleveland Clinic Score
Change from baseline in the severity of fecal incontinence | 3 Months
  The severity of fecal incontinence is evaluated using Cleveland Clinic Score
Change from baseline in the severity of fecal incontinence | 1 Month
  The severity of fecal incontinence is evaluated using Cleveland Clinic Score
Change from baseline on delay in postponing defecation | 6 Months
  postponing defecation delay is evaluated using a bowel diary
Change from baseline on delay in postponing defecation | 3 Months
  postponing defecation delay is evaluated using a bowel diary
Change from baseline on delay in postponing defecation | 1 Month
  postponing defecation delay is evaluated using a bowel diary
Change from baseline in the Number of active fecaI incontinence episodes per week | 6 months
  The number of fecaI incontinence episodes and/or urgencies is evaluated using a bowel diary
Change from baseline in the Number of active fecaI incontinence episodes per week | 3 months
  The number of fecaI incontinence episodes and/or urgencies is evaluated using a bowel diary
Change from baseline in the Number of urgencies episodes per week | 6 months
  The number of urgencies episodes is evaluated using a bowel diary
Change from baseline in the Number of urgencies episodes per week | 3 months
  The number of urgencies episodes is evaluated using a bowel diary

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie LEROI, Pr, Principal Investigator — University Hospital, Rouen
Locations (8):
- France (8):
  - Bordeaux University Hospital, Bordeaux
  - Clinique des Cèdres, Cornebarrieu
  - Hospices Civils de Lyon, Lyon
  - AP-HM Hôpital Nord, Marseille
  - AP-HP Hôpital Tenon, Paris
  - Hôpital des Diaconesses, Paris
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen

REFERENCES:
- [Derived] Leroi AM, Queralto M, Zerbib F, Siproudhis L, Vitton V, Amarenco G, Etienney I, Mion F, Bridoux V, Philip J, Brochard C, Damon H, Lacroix E, Gillibert A, Gourcerol G. Intrarectal injections of botulinum toxin versus placebo for the treatment of urge faecal incontinence in adults (FI-Toxin): a double-blind, multicentre, randomised, controlled phase 3 study. Lancet Gastroenterol Hepatol. 2024 Feb;9(2):147-158. doi: 10.1016/S2468-1253(23)00332-1. Epub 2023 Dec 18. PMID 38128556